CLINICAL TRIAL: NCT06646900
Title: Feasibility and Acceptability Trial of a Culturally Adapted Manual Versus Standard CBT Manual: A Randomized Control Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Association of Cognitive Therapists (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PACTMN24
Record Dates: First submitted 2024-06-14; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-06

CONDITIONS: Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: This will be a randomized controlled trial to evaluate the feasibility and acceptability of delivering a new intervention. Participants who meet the inclusion criteria will be randomly allocated to intervention or control groups in a 1:1 ratio.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- culturally adapted CaCBT manual (Experimental)
  Interventions: Behavioral: Culturally adapted CBT (CaCBT) based guided self-help manual
- standard CBT manual (Experimental)
  Interventions: Behavioral: Standard CBT Manual

INTERVENTIONS:
Behavioral: Culturally adapted CBT (CaCBT) based guided self-help manual — The intervention consists of seven modules including cognitive restructuring, problem solving, behavioural activation and conflict management. Three additional modules focus on interpersonal relationships, mental health wellbeing and self-care. Each module is delivered over one week. The intervention uses culturally appropriate stories, drawings, examples from local folklore and religious context to describe the concepts of CBT.
  Arms: culturally adapted CaCBT manual
Behavioral: Standard CBT Manual — The standard CBT manual will follow conventional CBT techniques without specific cultural adaptations
  Arms: standard CBT manual

SUMMARY:
This randomized controlled trial (RCT) will compare the efficacy and feasibility and acceptability of a culturally adapted CBT manual with a standard CBT manual, focusing on addressing cultural factors in therapy delivery.

DETAILED DESCRIPTION:
Randomized Controlled Trial (RCT): Participants will be randomly assigned to either the culturally adapted CBT manual group or the standard CBT manual group. A culturally adapted manual will integrate cultural values, norms, and idioms of suffering into CBT techniques, ensuring relevance and acceptance within the target cultural group. The standard CBT manual will follow conventional CBT techniques without specific cultural adaptations.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 18 to 65 years
2. 5 years of education
3. Symptoms of depression and anxiety

Exclusion Criteria:

1. Substance use disorder according to DSM-5 criteria as determined by primary care clinician
2. Significant cognitive impairment (for example, profound learning disability or dementia) as determined by primary care clinician
3. Active psychosis as determined by their primary care clinician

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2024-12-10 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility and acceptability measures | 12 weeks
  Feasibility and acceptability and Client's satisfaction will be measured through standardized measures of anxiety and depression
Clinical Measures | 12 weeks
  Depression and Anxiety, measured by Hosptal and Anxiety Scale (HADS)

CONTACTS AND LOCATIONS:
Locations (1):
- Pakistan Association of Cognitive Therapists, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No